CLINICAL TRIAL: NCT03785210
Title: Phase II Study of Nivolumab (Anti-PD1), Tadalafil and Oral Vancomycin in Patients With Refractory Primary Hepatocellular Carcinoma or Liver Dominant Metastatic Cancer From Colorectal or Pancreatic Cancers
Brief Title: Nivolumab (Anti-PD1), Tadalafil and Oral Vancomycin in People With Refractory Primary Hepatocellular Carcinoma or Liver Dominant Metastatic Cancer From Colorectal or Pancreatic Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190033; 19-C-0033
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Metastatic Pancreatic Cancer; Metastatic Colorectal Cancer; Liver Metastasis
Keywords: Anticancer Activities; Altering Gut Commensal Bacteria; Immunomdulatory Effect; Checkpoint Inhibition
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms | interventions — Nivolumab; Tadalafil; Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1 - Nivolumab, Tadalafil and Oral Vancomycin (Experimental): Nivolumab, tadalafil and oral vancomycin
  Interventions: Drug: nivolumab; Drug: tadalafil; Drug: oral vancomycin

INTERVENTIONS:
Drug: nivolumab — 480 mg intravenous (IV) every 4 weeks
  Other Names: Opdivo
Drug: tadalafil — 10 mg by mouth (PO) daily
  Other Names: Cialis
Drug: oral vancomycin — 125 mg every 6-hour (500 mg total daily dose) by mouth (PO) from week 1 to week 3, week 4 off.
  Other Names: Vancocin

SUMMARY:
Background:

A most common liver cancer in adults is hepatocellular carcinoma. Other kinds of liver cancer happen when colorectal or pancreatic cancer spreads to the liver. Researchers want to study if a combination of drugs helps people with these cancers. The drugs are nivolumab, tadalafil, and vancomycin.

Objective:

To investigate if nivolumab given with tadalafil and vancomycin causes liver cancer to shrink.

Eligibility:

Adults ages 18 years and older with hepatocellular carcinoma or metastases to the liver from colorectal or pancreatic cancer for which standard treatment has not worked

Design:

Participants will be screened with:

Medical and cancer history

Review of symptoms and ability to perform normal activities

Physical exam

Heart test. Some participants may meet with a cardiologist and/or have another heart test.

Scan of the chest, abdomen, and pelvis

Blood and urine tests

Tumor sample review. This can be from a previous procedure.

Participants will receive the study drugs in 4-week cycles. In each cycle participants will:

Get nivolumab through a small plastic tube in the arm on Day 1.

Take tadalafil by mouth 1 time every day.

Take vancomycin by mouth 4 times a day. They will take it every day for weeks 1 3, then not take it for week 4.

Complete a medicine diary of dates, times, missed doses and symptoms.

Throughout the study, participants will repeat screening tests and will give stool samples or rectal swabs.

After their last cycle, participants will have 3 follow-up visits over 3 months. Then they will be contacted every 6 months by phone or email and asked about their general well-being.

...

DETAILED DESCRIPTION:
Background:

* Current treatment options for patients with liver cancers, including hepatocellular carcinoma (HCC) and advanced liver cancers are limited and take no account of the known biological and genetic heterogeneity in these diseases. Median survival for advanced disease remains poor at approximately 1 year.
* Nivolumab is a fully human monoclonal immunoglobulin G4 (IgG4) antibody that is specific for human programmed death-1 (PD-1, cluster of differentiation 279 [CD279]) cell surface membrane receptor. Nivolumab has been approved by the Food and Drug Administration (FDA) for the treatment of HCC and other solid tumors.
* Tadalafil is a phosphodiesterase type 5 (PDE5) inhibitor which have been approved by the FDA for the treatment of pulmonary arterial hypertension, benign prostatic hyperplasia and erectile dysfunction, with a relative safe clinical profile. PDE5 inhibitors have been examined in multiple malignancies and cancer cell lines for their direct anticancer activities, for their

efficacy as chemo-sensitizers and for cancer chemoprevention.

* Oral vancomycin is antibiotic that has effect on altering gut commensal bacteria subsequently inducing a liver-selective anti-tumor effect.
* The aim of the study is to evaluate whether the immunomodulatory effect induced by PDE5 inhibitor and oral vancomycin can be enhanced by immune checkpoint inhibition in advanced liver cancer.

Objective:

-To determine the Best Overall Response (BOR) according to Response Evaluation Criteria (RECIST 1.1) to combined treatment of nivolumab, oral vancomycin and tadalafil in patients with refractory primary HCC or liver dominant metastatic cancer from colorectal cancer (CRC) or pancreatic adenocarcinoma (PDAC).

Eligibility:

* Histologically confirmed, hepatocellular carcinoma (HCC) Or
* Histologically confirmed carcinoma highly suggestive of a diagnosis of HCC Or
* Histologically confirmed advanced colorectal or pancreatic malignancy with liver involvement as dominant site of metastasis
* Measurable lesion, accessible for biopsy.
* Age greater than or equal to 18 years
* ECOG less than or equal to 1
* Acceptable renal, bone marrow and liver function.
* Willingness to undergo two mandatory tumor biopsies.

Design:

* The proposed study is a phase II study of combined nivolumab, oral vancomycin and tadalafil treatment in patients with HCC or liver dominant metastatic cancer from colorectal or pancreatic cancers.
* Treatment will be delivered in cycles consisting of 4 weeks (+/- 3 days) until progression or unacceptable toxicity.
* Patients will be seen in Clinical Center on monthly basis with disease status evaluation every

  8 (+/-1) weeks after start of study therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have

  * histopathological confirmation of Hepatocellular Carcinoma (HCC) (Cohort 1) OR
  * histopathological confirmation of carcinoma by in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC (Cohort 1) OR
  * histopathological confirmation of advanced colorectal or pancreatic malignancy with liver involvement as dominant site of metastasis (Per multidiscipline tumor board review and approval) (Cohort 2).
* Patients must have disease that is not amenable to potentially curative resection, transplantation or ablation.
* Patients must have progressed on, been intolerant to, or refused prior sorafenib/lenvatinib and/or atezolizumab/bevacizumab therapy (Cohort 1 only).
* Subjects must have progressed on or after standard systemic chemotherapy (at least one line of chemotherapy for patients with liver metastasis from pancreatic ductal adenocarcinoma (PDAC), at least two lines of chemotherapy for patients with liver metastasis from colorectal cancer (CRC) (Cohort 2 only).
* Patients must have evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Patients must have lesion accessible for biopsy and be willing to undergo pre- and posttreatment biopsies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* If liver cirrhosis is present, patient must have a Child-Pugh score less than or equal to 7
* Active chronic hepatitis B virus (HBV) infected subjects must be on antivirals and have HBV deoxyribonucleic acid (DNA) <100IU/mL. hepatitis C virus (HCV) infected subjects can be enrolled with close HCV RNA level monitoring.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of nivolumab in combination with tadalafil and vancomycin in patients less than 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Adequate hematological function defined by:

  * white blood cell (WBC) count greater than or equal to 3x10^9/L
  * absolute neutrophil count (ANC) greater than or equal to 1.5x10^9/L,
  * lymphocyte count greater than or equal to 0.5x10^9/L,
  * platelet count greater than or equal to 60x10^9/L, and
  * Hemoglobin (Hgb) greater than or equal to 9 g/ dL (more than 48 hours post-completion of blood transfusion)
* Adequate hepatic function defined by:

  * a total bilirubin level less than or equal to 1.5 X Upper limit of normal (ULN),
  * an aspartate transaminase (AST) level <5xULN,
  * an alanine aminotransferase (ALT) level <5xULN.
* Adequate renal function defined by:

  * Creatinine clearance (CrCl) greater than or equal to 50 mL/min/1.73 m^2 by 24 hours urine collection or as predicted by the Cockcroft-Gault formula:
  * CrCl = (140 age (y)) x (weight in kg) x (0.85, if female) x1.73 m^2/72 x Serum Creatinine (mg/dL) x patient's body surface area (BSA) (m^2) Or
* The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and up to 5 months (women) and 7 months (men) after the last dose of the drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patients with a history of cardiovascular disease may be enrolled per cardiology consultation and approval with echocardiogram and troponin level in normal range at the time of enrollment.
* Patient must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had standard-of-care anti-cancer therapy or therapy with investigational agents (e.g., chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigation agents), large field radiotherapy, or major surgery within 4 weeks prior to enrollment.
* Therapy with antibiotics within 30 days prior to enrollment.
* Therapy with nitrates, alpha-blockers, or cytochrome P450 (CYP3A4) inhibitors within 7- days prior to enrollment and for whom stopping is unsafe and/or a safe substitute is not medically recommended. Use of PDE5 inhibitors such as vardenafil (Levitra), tadalafil (Cialis), and sildenafil citrate (Viagra) less than or equal to 15-days prior to enrollment.
* The patient must not be currently on a corticosteroid dose greater than physiologic replacement dosing defined as 10 mg of cortisone per day or its equivalent.
* For PDAC patients with liver metastases, primary PDAC has not been resected (unless the primary is in the tail of the pancreas).
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Have signs of liver failure, e.g., clinical significant ascites, encephalopathy, or variceal bleeding within 6 months prior to enrollment.
* Prior major liver resection: remnant liver <50% of the initial liver volume. Patients with a biliary stent can be included.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or Chronic Inflammatory Demyelinating Polyneuropathy (CIDP), myasthenia gravis; systemic autoimmune disease such as Systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome. Such diseases should be excluded because of the risk of recurrence or exacerbation of disease.

Of note, patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.

* Have history of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with myocardial infarction or myocarditis within 12 months prior to enrollment.
* History of severe or unstable cerebrovascular disease.
* Sustained hypotension (<90/50 mmHg) or uncontrolled hypertension (>160/100 mmHg)
* Stroke within 6 months prior to enrollment.
* Human immunodeficiency virus (HIV)-positive patients are excluded because HIV causes complicated immune deficiency and study treatment can possess more risks for these patients.
* Have had prior transplant of any kind.
* Have ascites.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, tadalafil or vancomycin.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years prior to enrollment.
* Pregnant women are excluded from this study because nivolumabs potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, breastfeeding should be discontinued if the mother is treated with nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the Database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the Database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0033.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma: Participants with hepatocellular carcinoma highly suggestive of a diagnosis of hepatocellular carcinoma. Nivolumab 480 mg intravenously every 4 weeks; Tadalafil 10mg by mouth (PO) daily, and oral vancomycin 125mg every 6 hours by mouth (PO) from week 1 to week 3, week 4 off, 500 mg total daily.
- Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases: Participants with liver metastases from colorectal cancer or pancreatic ductal adenocarcinoma (PDAC). Nivolumab 480 mg intravenously every 4 weeks; Tadalafil 10mg by mouth (PO) daily, and oral vancomycin 125mg every 6 hours by mouth (PO) from week 1 to week 3, week 4 off, 500 mg total daily.
Period: Overall Study
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases
Started | 6 | 16
Completed | 5 | 10
Not Completed | 1 | 6
Not completed — Principal investigator decision - clinical progression | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 11 | 12
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.08 (8.15) | 63.61 (11.52) | 65.1 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 16 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 1 | 10 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 22

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR)
Description: Best overall response is defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started) assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Every 2 months and then every 6 months after discontinuation of treatment, for survival purposes, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases
Number analyzed (Participants) | 6 | 16
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 1 | 1
  Progressive Disease | 4 | 9
  Not Evaluable | 1 | 6

2. Secondary Outcome: Serious Adverse Events Possibly, Probably, and/or Definitely Related to Treatment
Description: Adverse events were assessed by the by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From first study treatment, approximately 90 days
Measure: Number; unit: adverse events
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases
Number analyzed (Participants) | 6 | 16
adverse events | 0 | 0

3. Secondary Outcome: Overall Survival (OS) of Nivolumab Combined With Oral Vancomycin and Tadalafil in Participants With Refractory Hepatocellular Carcinoma (HCC) or Liver Dominant Metastatic Cancer From Colorectal Cancer or Pancreatic Ductal Adenocarcinoma (PDAC)
Description: Overall survival is calculated from the on-study date to the day of death using the Kaplan-Meier method.
Time Frame: Participants were followed from the on-study date to post discontinuation of treatment until the day of death, an average of 8 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases
Number analyzed (Participants) | 6 | 16
Months | 9.4 [2.4 to 18.3] | 3.4 [2.6 to 8.7]

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 41 months/11 days and 36 months/22 days for the first and second group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases
Number analyzed (Participants) | 6 | 16
Participants | 6 | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 41 months/11 days and 36 months/22 days for the first and second group respectively.
Description: No deaths were related to research.
Arm/Group | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases
All-Cause Mortality (participants affected / at risk) | 5/6 | 15/16
Serious Adverse Events (participants affected / at risk) | 2/6 | 7/16
Other Adverse Events (participants affected / at risk) | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma (N=6) | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1, Arm 1, Treatment Assignment Code 1, Participants With Hepatocellular Carcinoma (N=6) | Cohort 2, Arm 1, Treatment Assignment Code 1, Participants With Liver Metastases (N=16)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 5 (6)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 3 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 4 (9)
Anemia (Blood and lymphatic system disorders) | 5 (7) | 12 (20)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 7 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 4 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 2 (2) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 2 (2) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 9 (9)
Fever (General disorders) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 9 (12)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 7 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 7 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 2 (5) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (7) | 9 (19)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, Altered mental status (Nervous system disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (3) | 4 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 4 (5) | 3 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Skin and subcutaneous tissue disorders - Other, blister right bottom foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03785210/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03785210/ICF_001.pdf